CLINICAL TRIAL: NCT03644407
Title: Galeazzi Spine Registry: Prospective Study for Clinical Monitoring of Patients Undergoing Spine Surgery
Brief Title: Galeazzi Spine Surgery RegistryGaleazzi Spine Registry: Prospective Study for Clinical Monitoring
Acronym: SPINEREG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: SPINEREG
Record Dates: First submitted 2018-04-25; First posted 2018-08-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Patients Undergoing Spine Surgery; Scoliosis; Disc Disease; Disc Injury; Myelopathy; Spinal Stenosis; SPINAL Fracture; Spinal Fusion
Keywords: registry; scoliosis; disc disease; spinal fracture; spinal fusion; spine surgery
MeSH Terms: conditions — Scoliosis; Spinal Cord Diseases; Spinal Stenosis; Spinal Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Spine Surgery — Patients undergoing spine surgery, who are the subjects eligible for participation to this observational prospective registry

SUMMARY:
The SPINEREG study is a prospective observational registry. Eligible patients are subjects undergoing spine surgery at the participating institutions.

Baseline health status and follow-up health status are recorded at pre-established steps.

DETAILED DESCRIPTION:
The SPINEREG study is a prospective observational study. Eligible patients are subjects undergoing spine surgery at the participating institutions.

Baseline health status and follow-up health status are recorded at pre-established steps.

Data from surgery and patients PROMs are registered on the database; the main timepoints are: pre-surgery, surgery, 3-6 month after surgery, 1-2-5-10-15-20 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spine surgery in the participating centers

Exclusion Criteria:

* Patients only in conservative treatment
* Patients to refuse to enter the study

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who undergo spine surgery in the participating centers and give informed consent to participate
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-11-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Spinal function (Oswestry Disability Index score) | 1 years
  Oswestry Disability Index score (ODI). Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Reliability of the data collected in SpineReg | 6 months
  This project was based on the retrospective analysis of patients prospectively enrolled in a spinal surgery registry, SpineREG. The study aims to evaluate the equivalence of the PROMs registered in SpineREG using two different formats: paper vs. electronic version. Through the comparison between the data electronically provided in SpineREG and the paper questionnaires, the accuracy, reliability and validity of the data were evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Briguglio M, Campagner A, Langella F, Cecchinato R, Damilano M, Bellosta-Lopez P, Crespi T, De Vecchi E, Latella M, Barone G, Scaramuzzo L, Bassani R, Luca A, Brayda-Bruno M, Wainwright TW, Middleton RG, Lombardi G, Cabitza F, Banfi G, Berjano P. Malnutrition and Disability: A Retrospective Study on 2258 Adult Patients Undergoing Elective Spine Surgery. Medicina (Kaunas). 2025 Feb 26;61(3):413. doi: 10.3390/medicina61030413. PMID 40142224
- [Derived] Bassani R, Morselli C, Cirullo A, Pezzi A, Peretti GM. A novel less invasive endoscopic-assisted procedure for complete reduction of low-and high-grade isthmic spondylolisthesis performed by anterior and posterior combined approach. Eur Spine J. 2023 Aug;32(8):2819-2827. doi: 10.1007/s00586-023-07666-9. Epub 2023 Mar 31. PMID 37000218